CLINICAL TRIAL: NCT05004350
Title: A Multicenter, Randomized, Open-label, 2-arm, Phase II Study With a Safety lead-in Phase Evaluating the Combination of Encorafenib and Cetuximab Versus Irinotecan/Cetuximab or Infusional 5-fluorouracil (5-FU)/Folinic Acid (FA)/Irinotecan (FOLFIRI)/Cetuximab in Chinese Patients With BRAF V600E Mutant Metastatic Colorectal Cancer.
Brief Title: A Study Evaluating the Combination of Encorafenib and Cetuximab Versus Irinotecan/Cetuximab or Infusional 5-fluorouracil (5-FU)/Folinic Acid (FA)/Irinotecan (FOLFIRI)/Cetuximab in Chinese Patients With BRAF V600E Mutant Metastatic Colorectal Cancer.
Acronym: NAUTICALCRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W00090GE202
Record Dates: First submitted 2021-04-30; First posted 2021-08-13 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: BRAF V600E; Metastatic Colorectal Cancer
Keywords: BRAF V600E; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — encorafenib; Cetuximab; IFL protocol; Leucovorin; Fluorouracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Encorafenib and cetuximab (Experimental): Safety Lead-in (SLI) phase:
  28 day cycles of encorafenib once daily (QD) 300 mg (4 x 75 mg oral capsule) and cetuximab 400 mg/m² initial dose (120-minute infusion), then 250 mg/m² (60-minute infusion) thereafter once weekly
  Randomized (Phase II) phase:
  28 day cycles of encorafenib once daily (QD) 300 mg (4 x 75 mg oral capsule) and cetuximab 400 mg/m² initial dose (120-minute infusion), then 250 mg/m² (60-minute infusion) thereafter once weekly
  Interventions: Drug: Encorafenib; Drug: Cetuximab
- Irinotecan and cetuximab or FOLFIRI and cetuximab (Experimental): Randomized (Phase II) phase: Either irinotecan and cetuximab or FOLFIRI and cetuximab in 28 day cycles.
  Irinotecan and cetuximab:
  * irinotecan 180 mg/m² (90-minute intravenous infusion or to study site standards) every 2 weeks and
  * cetuximab 400 mg/m² initial dose (120-minute intravenous infusion), then 250 mg/m² (60-minute infusion) thereafter once weekly
  OR
  FOLFIRI and cetuximab:
  * irinotecan 180 mg/m² (90-minute intravenous infusion or to study site standards) every 2 weeks
  * Folinic acid 400 mg/m² (120-minute infusion or to study site standards) or maximal dose tolerated in a prior regimen every 2 weeks
  * 5-FU 400 mg/m² initial dose bolus (not to exceed 15 minutes), then 1200 mg/m²/day × 2 days (total 2400 mg/m² over 46 to 48 hours) continuous infusion or maximal dose tolerated in a prior regimen every 2 weeks and
  * cetuximab 400 mg/m² initial dose (120-minute intravenous infusion), then 250 mg/m² (60-minute infusion) thereafter once weekly
  Interventions: Drug: Encorafenib; Drug: Cetuximab; Drug: FOLFIRI

INTERVENTIONS:
Drug: Encorafenib — oral hard capsule
  Other Names: Braftovi®; PF-07263896; W0090; LGX818; ONO-7702
Drug: Cetuximab — intravenous infusion
  Other Names: Erbitux®; C225
Drug: FOLFIRI — Combination of:
  irinotecan ( also known as: Camptosar, Camptothecin-11 and CPT-11) intravenous infusion, folinic acid (also known as: 5-formyl tetrahydrofolic acid and leucovorin) intravenous infusion, and 5-FU (also known as; fluorouracil) intravenous bolus/intravenous infusion
  Other Names: Folinic acid + Fluorouracil + Irinotecan
  Arms: Irinotecan and cetuximab or FOLFIRI and cetuximab

SUMMARY:
Encorafenib is currently being developed (with or without binimetinib), in combination with cetuximab, for the treatment of adult patients with B-RAF proto-oncogene, serine/threonine kinase V600E mutant (BRAF V600E) metastatic colorectal cancer (mCRC), who have received prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria for Molecular Prescreening:

The following inclusion criteria must be met for a participant to be eligible to undergo molecular tumor prescreening:

* Chinese male or female participant with age ≥18 years at the time of informed consent.
* Histologically- or cytologically-confirmed colorectal cancer (CRC) that is metastatic.
* Eligible to receive cetuximab per Chinese approved label with regard to tumor Rat Sarcoma Viral Oncogene Homologue (RAS) mutation status (i.e. approved for Rat Sarcoma Viral Oncogene Homologue Wild Type(RAS wt) status).
* Able to provide a sufficient amount of representative tumor specimen for central prospective laboratory testing of B-RAF Proto-oncogene, Serine/threonine Kinase (BRAF) mutation status and also retrospective RAS wt status and Microsatellite Instability (MSI) testing.

Inclusion Criteria for Treatment Period:

The following inclusion criteria must be met for a participant to be eligible for this study:

* Chinese male or female participant with age ≥18 years at time of informed consent.
* Histologically or cytologically confirmed CRC that is metastatic and unresectable at time of study entry (i.e. not suitable for complete surgical resection at screening).
* Presence of a BRAF V600E mutation in tumor tissue previously determined by a local assay at any time before screening or by the central laboratory.

NOTE: Other protocol defined Inclusion criteria may apply

Exclusion Criteria for Molecular Prescreening:

Participants meeting any of the following criteria are not eligible to undergo molecular tumor prescreening:

* Prior anti-Epidermal Growth Factor Receptor (anti-EGFR) treatment
* More than two prior regimens in the metastatic setting.
* Known contraindication to receive cetuximab or irinotecan at the planned dose according to the most recent cetuximab and irinotecan local label.
* Known history of Gilbert's syndrome or is known to have any of the following genotypes: uridine 5'-diphospho-glucuronosyltransferase (UGT)1A1*6/*6, UGT1A1*28/*28 or UGT1A1*6/*28.
* Leptomeningeal disease.

Exclusion Criteria for Treatment Period:

* Prior treatment with any Proto oncogene Serine/threonine-Protein Kinase (RAF) inhibitor, cetuximab, panitumumab or other EGFR inhibitors.
* Symptomatic brain metastasis.
* Leptomeningeal disease.
* Use of any herbal medications/supplements or any medications or foods that are moderate or strong inhibitors or inducers of cytochrome P450 (CYP)3A4/5 ≤1 week before the start of study intervention.
* Known history of acute or chronic pancreatitis within 6 months before the start of study intervention.

NOTE: Other protocol defined Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
Safety Lead-in Phase: Incidence of Dose Limiting Toxicities (DLTs) during the DLT-evaluation period (which is the first 28 days after the first dose of study intervention in the SLI) | Day 1 to Day 28
Randomized Phase 2: Progression-free Survival (PFS) by Blinded (to treatment received) Independent Central Review (BICR) | Day 1 through to study completion, approximately from 12 to 29 months
  Defined as the time from the date of randomization to the earliest documented disease progression as determined by BICR assessment per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1., or death due to any cause

SECONDARY OUTCOMES:
Safety Lead-in Phase: Type and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 | Informed consent through to study completion, approximately from 18 to 35 months
Safety Lead-in Phase: Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes from baseline of physical examinations | Day 1 through to study completion, approximately from 18 to 35 months
  Standard physical examinations on cardiovascular, respiratory, gastrointestinal, dermatological, ophthalmological and neurological systems will be performed and will be evaluated based on normal/abnormal and clinical significance observations. Number of participants with TEAEs related to abnormal or clinical significance observations to the physical examinations after the start of study drug will be reported.
Safety Lead-in Phase: Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes in vital signs from baseline of vital sign examinations. | Day 1 through to study completion, approximately from 18 to 35 months
  Clinically notable elevated values: Systolic blood pressure (BP): ≥ 160 mmHg and an increase ≥ 20 mmHg from baseline; Diastolic BP: ≥ 100 mmHg and an increase ≥ 15 mmHg from baseline; Heart rate : ≥ 120 beats/min (bpm) with increase from baseline of ≥ 15 bpm; Weight (kg) increase from baseline of ≥ 10%; Body temperature(°C) ≥ 37.5°C). Clinically notable low values: Systolic BP: ≤ 90 mmHg with decrease from baseline of ≥ 20 mmHg; Diastolic BP: ≤ 50 mmHg with decrease from baseline of ≥ 15 mmHg; Heart rate: ≤ 50 bpm with decrease from baseline of ≥ 15 bpm; Weight: ≥ 20% decrease from baseline; Body temperature [°C]: ≤ 36 °C. Number of participants with TEAEs related to notable changes to the vital signs after the start of study drug will be reported.
Safety Lead-in Phase: Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes from baseline of 12-lead electrocardiograms (ECGs) | Day 1 through to study completion, approximately from 18 to 35 months
  12-lead ECGs will be obtained using an internationally recognized 12-lead cardiograph. Clinically notable ECG values: QT (ms) and QT interval (ms) corrected for heart rate using Fridericia's formula (QTcF) intervals (ms) : increase from baseline > 30 ms; increase from baseline > 60 ms, new > 450 ms, new > 480 ms, new > 500 ms. Heart rate (beats/min) : increase from baseline > 25% to a value > 100 bpm, decrease from baseline > 25% and to a value < 50 bpm. Number of participants with TEAEs related to abnormal or notable changes to ECG parameters after the start of study drug will be reported.
Safety Lead-in Phase: Incidence of treatment-emergent adverse events (TEAEs) related to notable changes in clinical safety laboratory parameters from baseline. | Day 1 through to study completion, approximately from 18 to 35 months
  Number of participants with clinically notable shift from baseline in laboratory parameter values based on national cancer institute common terminology criteria (NCI-CTCAE) grade, Version 4.03 were graded from Grades 1 to 5. Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local or noninvasive intervention indicated. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death. Clinically notable shift is defined as a worsening from baseline by at least 2 grades, or to grade 3 or above.
Safety Lead-in Phase: Incidence of development of of keratoacanthoma and/or squamous cell carcinoma and new primary melanoma by dermatological examinations | Screening (Day -28 to -1) through to study completion, approximately from 18 to 35 months
  This is to monitor for the possible development of keratoacanthoma and/or squamous cell carcinoma and new primary melanoma, as these have been reported to occur with selective BRAF inhibitor treatment. This assessment will be performed at screening and every 8 weeks from Cycle 1 Day 1 (i.e. on Day 1 of Cycles 1, 3, 5, 7…), the end of treatment visit and the 30-day safety follow up visit.
Safety Lead-in Phase: Performance status assessment using the Eastern Co-operative Oncology Group (ECOG) performance status scale | Screening (Day -28 to -1) through to study completion, approximately from 18 to 35 months
  Scale with a range from 0 to 5 with lower score mean a lower functional impairment, 5 corresponding to death
Safety Lead-in Phase: Incidence of dose interruptions, dose modifications and discontinuations due to adverse events (AEs) | Day 1 until end of treatment, approximately 1 year
Safety Lead-in Phase: Plasma concentrations of encorafenib | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Safety Lead-in Phase: Serum concentrations of cetuximab | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Safety Lead-in Phase; Pharmacokinetic (PK) parameter derived from plasma concentration of encorafenib area under curve (AUC) in Chinese participants | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Safety Lead-in Phase: Pharmacokinetic (PK) parameter derived from serum concentration of cetuximab area under curve (AUC) in Chinese participants | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Safety Lead-in Phase: Pharmacokinetic (PK) parameter derived from plasma concentration of encorafenib minimum concentration (Cmin) in Chinese participants | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Safety Lead-in Phase: Pharmacokinetic (PK) parameter derived from serum concentration of cetuximab minimum concentration (Cmin) in Chinese participants | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Safety Lead-in Phase: Pharmacokinetic (PK) parameter derived from plasma concentration of encorafenib maximum concentration (Cmax) in Chinese participants | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Safety Lead-in Phase: Pharmacokinetic (PK) parameter derived from serum concentration of cetuximab maximum concentration (Cmax) in Chinese participants | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Safety Lead-in Phase: Objective response rate (ORR) | Day 1 through to study completion, approximately from 18 to 35 months
  Objective response rate (ORR) defined as the proportion of participants with a best overall best response of either complete response (CR) or partial response (PR) as determined by Blinded (to treatment received) Independent Central Review (BICR) and investigator assessment per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Safety Lead-in Phase: Duration of Response (DOR) (months); defined for responders complete response (CR) or partial response (PR) only, is duration of time from the date of the first documented response to the earliest date of disease progression | Day 1 through to study completion, approximately from 18 to 35 months
  Duration of response, defined as the time from first documented response (complete response or partial response) to the earliest date of disease progression as determined by Blinded (to treatment received) Independent Central Review (BICR) and investigator assessment per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, or death due to underlying disease.
Randomized Phase 2: Progression-free survival (PFS) | Day 1 through to study completion, approximately from 12 to 29 months
  Progression-free survival defined as the interval of time between the date of randomization to the earliest date of disease progression, as determined by investigator assessment per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death due to any cause.
Randomized Phase 2: Overall Response Rate (ORR) | Day 1 through to study completion, approximately from 12 to 29 months
  Overall response rate (for confirmed and unconfirmed responses) defined as the proportion of participants with a confirmed (resp. unconfirmed) best overall response of either complete response or partial response, as determined by Blinded (to treatment received) Independent Central Review (BICR) and investigator assessment per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Randomized Phase 2: Duration of Response (DOR) | Day 1 through to study completion, approximately from 12 to 29 months
  Duration of response defined as the time from the date of the first documented response (complete response or partial response) to the earliest date of disease progression, as determined by Blinded (to treatment received) Independent Central Review (BICR) and investigator assessment per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death due to any cause
Randomized Phase 2: Disease control rate (DCR) | Day 1 through to study completion, approximately from 12 to 29 months
  Disease control rate (DCR), defined as the proportion of participants with a best overall response of either complete response, partial response or stable disease (SD), as determined by Blinded (to treatment received) Independent Central Review (BICR) and investigator assessment per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Randomized Phase 2: Time to Response (TTR) | Day 1 through to study completion, approximately from 12 to 29 months
  Time to Response (for confirmed and unconfirmed responses) is defined as the time between date of randomization until first documented response of complete response (CR) or partial response (PR).
Randomized Phase 2: Overall Survival (OS) | Day 1 through to study completion, approximately from 12 to 29 months
  Overall survival is defined as time from randomization until date of death due to any cause
Randomized Phase 2: Type and severity of adverse events (AEs) and serious adverse events (SAEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 | Informed consent date through to study completion, approximately from 12 to 29 months
Randomized Phase 2: Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes from baseline of physical examinations | Day 1 through to study completion, approximately from 12 to 29 months
  Standard physical examinations on cardiovascular, respiratory, gastrointestinal, dermatological, ophthalmological and neurological systems will be performed and will be evaluated based on normal/abnormal and clinical significance observations. Number of participants with TEAEs related to abnormal or clinical significance observations to the physical examinations after the start of study drug will be reported
Randomized Phase 2: Incidence of treatment-emergent adverse events (TEAEs) related to notable changes in vital signs from baseline. | Day 1 through to study completion, approximately from 12 to 29 months
  Clinically notable elevated values: Systolic blood pressure (BP): ≥ 160 mmHg and an increase ≥ 20 mmHg from baseline; Diastolic BP: ≥ 100 mmHg and an increase ≥ 15 mmHg from baseline; Heart rate : ≥ 120 beats/min (bpm) with increase from baseline of ≥ 15 bpm; Weight (kg) increase from baseline of ≥ 10%; Body temperature(°C) ≥ 37.5°C). Clinically notable low values: Systolic BP: ≤ 90 mmHg with decrease from baseline of ≥ 20 mmHg; Diastolic BP: ≤ 50 mmHg with decrease from baseline of ≥ 15 mmHg; Heart rate: ≤ 50 bpm with decrease from baseline of ≥ 15 bpm; Weight: ≥ 20% decrease from baseline; Body temperature [°C]: ≤ 36 °C. Number of participants with TEAEs related to notable changes to the vital signs after the start of study drug will be reported.
Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes to electrocardiogram evaluations from baseline | Day 1 through to study completion, approximately from 12 to 29 months
  12-lead ECGs will be obtained using an internationally recognized 12-lead cardiograph. Clinically notable ECG values: QT (ms) and QT interval (ms) corrected for heart rate using Fridericia's formula (QTcF) intervals (ms): increase from baseline > 30 ms; increase from baseline > 60 ms, new > 450 ms, new > 480 ms, new > 500 ms; Heart rate (beats/min): increase from baseline > 25% to a value > 100 bpm, decrease from baseline > 25% and to a value < 50 bpm. Number of participants with TEAEs related to abnormal or notable changes to ECG parameters after the start of study drug will be reported.
Randomized Phase 2: Incidence of treatment-emergent adverse events (TEAEs) related to notable changes in clinical safety laboratory parameters from baseline. | Day 1 through to study completion, approximately from 12 to 29 months
  Number of participants with clinically notable shift from baseline in laboratory parameter values based on national cancer institute common terminology criteria (NCI-CTCAE) grade, Version 4.03 were graded from Grades 1 to 5. Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local or noninvasive intervention indicated. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death. Clinically notable shift is defined as a worsening from baseline by at least 2 grades, or to grade 3 or above.
Randomized Phase 2: Incidence of development of keratoacanthoma and/or squamous cell carcinoma and new primary melanoma by dermatological examinations | Day 1 through to study completion, approximately from 12 to 29 months
  This is to monitor for the possible development of keratoacanthoma and/or squamous cell carcinoma and new primary melanoma, as these have been reported to occur with selective BRAF inhibitor treatment. This assessment will be performed at screening and every 8 weeks from Cycle 1 Day 1 (i.e. on Day 1 of Cycles 1, 3, 5, 7…), the end of treatment visit and the 30-day safety follow up visit.
Randomized Phase 2: To determine the performance status using the Eastern Co-operative Oncology Group (ECOG) performance status scale. | Day 1 through to study completion, approximately from 12 to 29 months
  Scale with a range from 0 to 5 with lower score mean a lower functional impairment, 5 corresponding to death
Randomized Phase 2: To determine if there is any change from baseline in the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer Patients (EORTC QLQ-C30) questionnaire scores | Day 1 through to study completion, approximately from 12 to 29 months
  EORTC QLQ-C30 consist of nine multi-item scales: five functional scales (physical, role, cognitive, emotional and social); three symptom scales (fatigue, pain, nausea and vomiting); and a global health and Quality of Life (QoL) scale. Each scale in the questionnaire will be scored (0 to 100). High scores represents a high health/quality of life
Randomized Phase 2: To determine if there is any change from baseline in the European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) questionnaire scores. | Day 1 through to study completion, approximately from 12 to 29 months
  EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (VAS). The descriptive system has five dimension (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), each is rated according to a five-point verbal rating scale (VRS): 1. no problems, 2. slight problems, 3. moderate problems, 4. severe problems and 5. extreme problems) and translated into a five-digit number that describes the participant's health state.
Randomized Phase 2: To determine if there is any change from baseline in the Functional Assessment of Cancer Therapy-Colon Cancer (FACT-C) questionnaire scores | Day 1 through to study completion, approximately from 12 to 29 months
  FACT-C is a validated quality of life questionnaire for patient reported outcome assessment. FACT-C consists of 36 items, presented on a five-point Likert scale, in four domains of well-being (physical, emotional, social and functional) and the Colorectal Cancer Subscale. Higher score reflects a better quality of life.
Randomized Phase 2: To determine if there is any changes in the Patient Global Impression of Change (PGIC) questionnaire scores. | Day 1 through to study completion, approximately from 12 to 29 months
  PGIC will ask participants to evaluate their CRC symptoms since starting study intervention according to a seven-point verbal rating scale (VRS): 1. very much improved, 2. much improved, 3. minimally improved, 4. no change, 5. minimally worse, 6. much worse, 7. very much worse
Randomized Phase 2: Plasma concentrations of encorafenib | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Randomized Phase 2: Serum concentrations of cetuximab | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Randomized Phase 2; Pharmacokinetic (PK) parameter derived from plasma concentration of encorafenib area under curve (AUC) in Chinese participants | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Randomized Phase 2: Pharmacokinetic (PK) parameter derived from serum concentration of cetuximab area under curve (AUC) in Chinese participants | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Randomized Phase 2: Pharmacokinetic (PK) parameter derived from plasma concentration of encorafenib minimum concentration (Cmin) in Chinese participants | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Randomized Phase 2: Pharmacokinetic (PK) parameter derived from serum concentration of cetuximab minimum concentration (Cmin) in Chinese participants | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Randomized Phase 2: Pharmacokinetic (PK) parameter derived from plasma concentration of encorafenib maximum concentration (Cmax) in Chinese participants | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Randomized Phase 2: Pharmacokinetic (PK) parameter derived from serum concentration of cetuximab maximum concentration (Cmax) in Chinese participants | Day 1 of Cycles 1 and 2; Each cycle = 28 days
Randomized Phase 2: Population pharmacokinetic (PK) analysis using the ARRAY 818 302 study PK data | Day 1 through to study completion, approximately from 12 to 29 months

OTHER OUTCOMES:
Randomized Phase 2: Changes from baseline in blood Carcinoembryonic Antigen (CEA) and Cancer Antigen 19-9 (CA19-9) at the beginning of each cycle and at the end of treatment | Screening (Day -28 to -1) through to study completion, approximately from 12 to 29 months
Randomized Phase 2: Microsatellite Instability (MSI) status in Formalin-fixed and Paraffin Embedded (FFPE) samples using established Polymerase Chain Reaction (PCR) assays in tumor sample versus germline control at screening | Screening (Day -28 to Day -1)

CONTACTS AND LOCATIONS:
Overall Officials: Shen Lin, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (34):
- China (34):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Medical University - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital Sun Yat-Sen University, Guangzhou, Guangdong
  - Cancer Hospital Affiliated to Shantou University Medical College, Shantou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Affiliated Hospital of Hebei University, Baoding, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji medical college Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affilliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Tongji University, Shanghai, Shanghai Municipality
  - The Second People's Hospital of Neijiang, Neijiang, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital - Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital - Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No